CLINICAL TRIAL: NCT04678245
Title: Testing Peer-led Network Intervention to Prevent Adolescent Vaping
Brief Title: Network Intervention to Prevent Vaping
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Texas Tech University (Other); Claremont Graduate University (Other); Penn State University (Other); University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Peter A. Wyman, Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R01DA050991 (NIH); 1R01DA050991 (NIH)
Record Dates: First submitted 2020-04-02; First posted 2020-12-21 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Vaping; Preventive Psychiatry; Social Networking
Keywords: preventive intervention; e-cigarettes; middle school; high school; messaging; network informed prevention
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Intervention Model Description: Immediate intervention and delayed intervention groups - by school over 2 cohorts
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate Above the Influence-Vaping Intervention (Experimental): School receives Above the Influence-Vaping (ATI-V) prevention program training after baseline assessment. Training and intervention continue over two school years (approximately 18 months). Surveys at baseline, 8 months (end 8th grade), 20 mo (end 9th grade), 28 mo (mid-10th grade).
  Interventions: Behavioral: Above the Influence-Vaping (ATI-V)
- Delayed Above the Influence-Vaping Intervention (Active Comparator): Surveys at baseline, 8 months (end 8th grade), 20 mo (end 9th grade), 28 mo (mid-10th grade). ATI-V prevention program training after 4th assessment - after 28 months.
  Interventions: Behavioral: Above the Influence-Vaping (ATI-V)

INTERVENTIONS:
Behavioral: Above the Influence-Vaping (ATI-V) — Peer-nominated 8th grade and 9th grade Peer Leaders (PL) will be trained in a half day ATI-V training. Adult Advisors (AA) will attend a half day ATI-V AA training and the PL training. The training day builds leadership skills in the PLs, develops skills for rising above pressure to vape including identification of personal reasons to rise, identification of healthy support people, teaching accurate use statistics, and sharing stories of prior success in rising above negative pressures. The ATI-V team of PLs and AAs then will run four interactive messaging campaigns to reach the rest of the student body. These four campaigns are (1) Introduction to ATI-V and My Reasons to Rise (2) Gain and Loss (3) Who's Got My Back (4) The Facts. Each campaign features a portion in which PLs model healthy norms and behaviors, and a second portion in which all the rest of the students engage in an interactive component to build and demonstrate the target skill.

SUMMARY:
Rates of adolescent vaping are increasing rapidly. Current high school student use of electronic vaping products (EVPs) rose from 1.5% in 2011 to 20.8% in 2018 - an increase from 220,000 to 3.05 million adolescent users. Effective, school-based interventions are urgently needed to protect adolescents from initiating or continuing use of electronic vaping products (EVPs). This study leverages a state-supported prevention initiative to test the effectiveness of a promising intervention that trains 8th-9th grade student peer leaders to deliver school-wide vaping prevention campaigns with ongoing adult mentoring. If study hypotheses are supported, the study will provide the first evidence of a school-based preventive intervention that reduces adolescent vaping behaviors, as well as insight into how peer communications can be harnessed to prevent vaping.

DETAILED DESCRIPTION:
Above the Influence of Vaping (ATI-V) trains peer nominated 8th-9th grade Peer Leader, and adult advisors. Peer Leaders learn skills and implement school-wide prevention campaigns informed by communication science.New York State has provided funds to support schools to implement ATI-V but no funds for efficacy research. With support from New York State and a strong team of investigators, our project has two aims:

Aim 1. Efficacy. The primary aim of this study is to determine ATI-V impact in preventing vaping use (past 30 days any vaping, nicotine vaping, and regular use). Using an RCT design, 20 schools will be assigned to (a) immediate ATI-V, or (b) wait-list for ATI-V training after 24 months. Approximately 3,800 8th graders will be enrolled and followed for assessments in fall 8th grade, spring 8th grade, spring 9th grade, and mid-year 10th grade. We will test for which students ATI-V is most effective and in what school contexts (school climate).

Aim 2. Mechanism. The second aim of this study to test the hypothesized mechanisms of ATI-V impact. To accomplish this aim we will conduct statistical analyses of a mediation model to determine (a) whether ATI-V improves students' perceptions that vaping is unacceptable to their peers (anti-vaping norms), connections to supportive adults to address EVP concerns, and social influence of non-vaping students; and (b) whether the impact of ATI-V on reduced vaping behavior is mediated by these improvements.

ELIGIBILITY:
Inclusion Criteria:

* current 8th grade student of study school at start of school participation
* No person shall be excluded from participation, denied benefits, or discriminated against because of race, color, national origin, sexual orientation, sex, gender identity, age, or ability (i.e., special education status).

Exclusion Criteria:

* non-English speaking students

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 3840 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-10-04 (Estimated)

PRIMARY OUTCOMES:
Number of participants with any past 30 day any vaping | 28 months
  Self-report of e-cigarette use of any kind in the past 30 days (Johnston, et al., 2019)
Number of participants with any past 30 day nicotine vaping | 28 months
  self-report of e-cigarette use with nicotine product in the past 30 days (Johnston, et al., 2019)

SECONDARY OUTCOMES:
Score Electronic Vaping Product Harm | 28 months
  self report of 'how much do you think people risk harming themselves (physically or in other ways) when they use electronic vapor products every day?' on a 4 point likert scale of No risk (0) to Great risk (3) (Johnston, et al., 2019) Higher numbers suggest perception of greater harm. This one item scale will range from 0 to 3.
Mean Electronic Vaping Product Attitudes | 28 months
  mean of self report items of whether vaping is 'good, fun, interesting, exciting' on a 5 point likert scale of Strongly disagree (1) to Strongly agree (5) (Ajzen, 2001). Higher numbers suggest more positive attitudes towards vaping. Scale is mean, so will range from 1 to 5.
Total Number of Trusted Adults | 28 months
  self report of adults at school students can 'trust or feel you can talk to about personal things'. Can name up to 7 adults - reporting total number (range 0-7).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data (stripped of school names and other identifiers) for all primary and secondary outcome measures will be made available to collaborators and other interested researchers via secure server links.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be available within 6 months of study completion.
Access Criteria: Requestors will be required to sign a data access agreement. The data sharing agreement involves sharing only de-identified data with other investigators and the use of data sharing agreements that provide for: (1) a commitment for using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed.

REFERENCES:
- [Background] Ajzen I. Nature and operation of attitudes. Annu Rev Psychol. 2001;52:27-58. doi: 10.1146/annurev.psych.52.1.27. PMID 11148298
- [Background] Johnston, L. D., Miech, R. A., O'Malley, P. M., Bachman, J. G., Schulenberg, J. E., & Patrick, M. E. (2019). Monitoring the Future National Survey Results on Drug Use, 1975-2018: Overview, Key Findings on Adolescent Drug Use. Institute for Social Research.
- [Background] Wyman PA, Pickering TA, Pisani AR, Rulison K, Schmeelk-Cone K, Hartley C, Gould M, Caine ED, LoMurray M, Brown CH, Valente TW. Peer-adult network structure and suicide attempts in 38 high schools: implications for network-informed suicide prevention. J Child Psychol Psychiatry. 2019 Oct;60(10):1065-1075. doi: 10.1111/jcpp.13102. Epub 2019 Aug 8. PMID 31392720